CLINICAL TRIAL: NCT04490447
Title: Identification of Microbiome and Metabolome of Bronchiectasis in Chinese Population and Role of the "Gut-lung Axis" in Chronic Respiratory Infection With Pseudomonas Aeruginosa.
Brief Title: Identification of Microbiome and Metabolome of Bronchiectasis in Chinese Population.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Director, Head of respiratory medicine, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 20190403
Record Dates: First submitted 2020-04-24; First posted 2020-07-29 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — faecal samples for 16S rRNA sequencing and LC-MS analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bronchiectasis: Patient meets diagnose of bronchiectasis refering to "BTS guideline 2010" will be included.
- Healthy control: Healthy volunteers will be included.

SUMMARY:
This study aims to investigate the characteristics of gut microbiome and metabolome in non-CF bronchiectasis patients, hoping to explore the underlying mechanisms as well as the influence of gut microbiota composition on bronchiectasis.

DETAILED DESCRIPTION:
Non-cystic fibrosis bronchiectasis is a chronic airway disease characterized by irreversible and progressive dilation of the large airways, bronchi and bronchioles, which severely impairs the life quality of patients and increases the social and economic burden. It is also a heterogenous disease affected by multiple factors such as geography and ethnicity. The incidence of bronchiectasis among the Chinese population is about 1.2%, which has clearly been underestimated. However, due to the lack of awareness, the research of bronchiectasis in China is still in its infancy. Colonization and recurrent infection of pathogen is the primary unsolved problem in clinical practice. With the proposition of "gut-lung axis" theory, the role of gut microbiota in the pathogenesis of respiratory diseases has been gradually revealed. Evidences have shown that gut microbiota regulates respiratory immunity via releasing soluble bacterial components and its metabolites into the circulation, as well as facilitating the migration of immune cells directly to the lung. In the 1980s, a patient after a colectomy has been reported to generate bronchiectasis. The most common clinical manifestation of pulmonary involved IBD patients is also bronchiectasis, suggesting that the "gut-lung axis" may be involved in the pathogenesis of bronchiectasis. Therefore, clarifying the role and mechanism of gut microbiota in bronchiectasis and its gut microbiome is expected to provide new theoretical basis and ideas for its diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Regular bowel movement: every 2 days - 3 times/ day
* The diagnose of bronchiectasis should refer to "BTS guideline 2010"

Exclusion Criteria:

* Diagnosis of ABPA
* Pregnancy or lactation
* Active smoking or alcohol using within last 6 months
* HIV infection
* Previous abdominal or rectal surgery
* Diagnosis of chronic gastrointestinal disease, heart disease, diabetes, severe renal insufficiency (GFR < 30ml/min) or immunodeficiency
* Regular use of the following types of medications (> 2 times per week) within last 2 months: opium, loperamide antidiarrheal, systemic antihistaminic, metoclopramide, proton pump inhibitor
* Poor compliance or inability to cooperate as judged by the doctor

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled in this study should meet the diagnositc criteria of BTS guideline 2010" . Patients with a history of antibiotic use were admitted to the study. Healthy volunteers were eligible for inclusion provided they had not received antibiotics within the previous one month.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-06-22 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome and metabolomics of bronchiectasis patients and healthy control. | 12 months
  The microbiome and metabolome results of gut in bronchiectasis patients will be defined from the stool samples using 16S rRNA Miseq sequencing and nontargeted LC-MS-based metabolomics approach.

SECONDARY OUTCOMES:
Lung microbiome of bronchiectasis patient. | 12 months
  The bronchoalveolar lavage fluid (BALF) specimens will be obtained from admitted patients undergoing bronchoscopy and the lung microbiome of bronchiectasis patients will be defined from the BALF samples using 16S rRNA Miseq sequencing.
BSI (Bronchiectasis Severity Index) score | 2 months
  Assessment of the non-cystic fibrosis bronchiectasis severity according to the BSI score at the time of enrollment.
  BSI score: scale of 0-26, is calculated from the results of age, BMI(body mass index), FEV1% predicted, exacerbations, hospital admissions, airway organisms colonisation, radiological severity etc.) 0-4, 5-8, >9 were separately defined as mild, moderate, severe bronchiectasis, higher score indicates probable higher mortality rate and hospitalisation rate.
Lung function | 12 months
  Lung function will be accessed by Pulmonary Function Tests (PFT) and the parameters including FVC ( forced vital capacity), FEV1 (forced the first second of expiratory volume), FEV1% predicted, FEV1/FVC will be documented at the time of enrollment
Sputum bacteriological evaluation. | 12 months
  Sputum bacteriological (pseudomonas aeruginosa and other organisms) will be evaluated.
Chest high-resolution computed tomography (CT). | 12 months
  Chest high-resolution computed tomography (CT) results in the recent 6 months will be documented.
Acute exacerbation | 12 months
  The time of acute exacerbation in the following year will be recorded according to medical information.
Hospitalization | 12 months
  The time of hospitalization in the following year will be recorded according to medical information.
Duration to the first exacerbation during the one-year follow up. | 24 months
  The duration to the first exacerbation within one year after the sample collection.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-fu Xu, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital , Tongji University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang WW, Mao B, Liu Y, Gu SY, Lu HW, Bai JW, Liang S, Yang JW, Li JX, Su X, Hu HY, Wang C, Xu JF. Altered fecal microbiome and metabolome in adult patients with non-cystic fibrosis bronchiectasis. Respir Res. 2022 Nov 19;23(1):317. doi: 10.1186/s12931-022-02229-w. PMID 36403022